CLINICAL TRIAL: NCT04093921
Title: Ready for Change: a Telehealth, Motivational Enhancement Pre-habilitation Training to Increase Engagement in Children and Families Entering Intensive Interdisciplinary Pain Rehabilitation
Brief Title: Ready for Change: Enhancing Motivational Engagement Prior to IIPT
Acronym: PREPaRe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Deirdre Logan, Director of psychology services in pain medicine, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P00033150
Record Dates: First submitted 2019-09-10; First posted 2019-09-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain
Keywords: chronic pain; pediatric
MeSH Terms: conditions — Chronic Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Those providing care at the PPRC will not know which study arm their patients were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Receive motivational enhancement training based, telehealth-delivered 6-8 session intervention aimed at increasing readiness to engage in pain self-management, in addition to all recommended outpatient treatments.
  Interventions: Behavioral: MET-based therapy; Behavioral: Standard Care
- Standard Care (Active Comparator): Participate in all recommended outpatient pain treatments while awaiting PPRC admission.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: MET-based therapy — see previous
  Arms: Intervention
Behavioral: Standard Care — To include all recommended outpatient treatments

SUMMARY:
This is a randomized, motivational-interviewing-based intervention to improve readiness-to-change, or willingness to engage in a self-management approach to chronic pain, for patients referred to our intensive interdisciplinary pain rehabilitation day program.

DETAILED DESCRIPTION:
Readiness to change, or willingness to engage in a self-management approach to chronic pain and disability, is the most powerful predictor of children's success in intensive pediatric pain rehabilitation. Motivational Enhancement Therapy (MET) is an approach that has been effective in increasing readiness to change and treatment engagement for other behaviorally-oriented health interventions. However, MET has never been systemically employed in the context of treating pediatric chronic pain and disability.

This demonstration project seeks to test the effects of a novel telehealth intervention using motivation enhancement therapy to improve patient and parent engagement in, and outcomes of, an intensive interdisciplinary day hospital program for children with complex chronic pain conditions and associated disability, the Pediatric Pain Rehabilitation Center (PPRC). The intervention, PPRC-Prep, is a 4 week MET-based telehealth intervention that will be offered to families of children with refractory chronic pain conditions awaiting admission to the PPRC at Boston Children's Hospital at Waltham. Families approved for and awaiting PPRC admission will be randomized to receive PPRC-Prep along with usual care or to a comparison group receiving treatment as usual. Study aims include assessing the feasibility and acceptability of the intervention along with measuring its potential to increase readiness to engage in a self-management approach assessed at time of admission to the PPRC using established measures of readiness to change, pain acceptance, and committed action. Investigators will also evaluate the effects of PPRC-Prep on program length of stay and on reductions of disability and pain at PPRC discharge and short-term (8-week) follow up through comparison of families who undergo PPRC-prep with families who do not undergo PPRC-prep. Demonstrating the feasibility and preliminary effectiveness of PPRC-Prep will enable the study team to establish this as a routine component of our approach to care for children with complex, refractory chronic pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 8-18 at enrollment
* Presence of chronic pain condition for > 3 months with moderate or severe disability
* Accepts referral to PPRC and awaiting admission

Exclusion Criteria:

* Non-English speaking
* No access to device with telehealth capability

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Length of stay | PPRC discharge [within 6 months of baseline]
  length of stay in PPRC program (in weeks)
Functional disability inventory (FDI) total score | at PPRC follow up (4-8 weeks post discharge)
  level of pain related functional disability, ranges from 0-60 with higher scores indicating more disability
Pain stages of change questionnaire for adolescents (PSOCQ-A) | PPRC admission (within 2 months of baseline)
  readiness to change/embrace pain self-management. 13 item scale with total scores ranging from 13-65. Domain with highest score is considered current stage of change.
Pain stages of change questionnaire for adolescents (PSOCQ-A) | PPRC discharge [within 6 months of baseline]
  readiness to change/embrace pain self-management. 13 item scale with total scores ranging from 13-65. Domain with highest score is considered current stage of change.
Pain stages of change questionnaire for adolescents (PSOCQ-A) | at PPRC follow up (4-8 weeks post discharge)
  readiness to change/embrace pain self-management. 13 item scale with total scores ranging from 13-65. Domain with highest score is considered current stage of change.
Pain stages of change questionnaire for adolescents (PSOCQ-A) | at PPRC follow up (1 year post discharge)
  readiness to change/embrace pain self-management. 13 item scale with total scores ranging from 13-65. Domain with highest score is considered current stage of change.
Modified Adolescent Treatment Engagement Questionnaire | At end of intervention, 4 weeks from baseline
  Level of engagement in treatment. Scores 0-40 higher scores indicate more engagement.
Chronic Pain Acceptance Questionnaire total score | At PPRC discharge [within 6 months of baseline]
  Measure of readiness to change/engage in pain self-management. 20 item questionnaire, will use total score. Range 0-120. HIgher scores indicate more pain acceptance.
Chronic Pain Acceptance Questionnaire total score | At PPRC admission [typically within 3 months of baseline]
  Measure of readiness to change/engage in pain self-management. 20 item questionnaire, will use total score. Range 0-120. HIgher scores indicate more pain acceptance.
Treatment satisfaction inventory | At end of intervention, 4 weeks from baseline
  Participant satisfaction with treatment. 13 items range 13-65, higher scores = more satisfaction
Readiness Rulers | During and at end of the intervention, for the treatment group only
  Motivational interviewing based ratings of willingness, importance, awareness and confidence related to adopting a self-management approach to pain

SECONDARY OUTCOMES:
Pain intensity | At PPRC admission (4-6 weeks post baseline)
  pain intensity on 0-10 numeric scale (10=worst pain)
Pain intensity | At PPRC discharge [within 6 months of baseline]
  pain intensity on 0-10 numeric scale (10=worst pain)
Functional disability inventory (FDI) total score | at PPRC discharge [within 6 months of baseline]
  level of pain related functional disability, ranges from 0-60 with higher scores indicating more disability
Functional disability inventory (FDI) total score | at PPRC follow up (1 year post discharge)
  level of pain related functional disability, ranges from 0-60 with higher scores indicating more disability
Pain intensity | At first post-treatment follow up (4-8 weeks post discharge)
  pain intensity on 0-10 numeric scale (10=worst pain)
Pain intensity | 1 year post-treatment
  pain intensity on 0-10 numeric scale (10=worst pain)
Committed action questionnaire total score | At PPRC admission [typically within 3 months of baseline]
  Secondary measure of readiness to change/engage in pain self-management. 8 item questionnaire with range 0-48. Higher scores indicate more committed action.
Committed action questionnaire | At PPRC discharge [within 6 months of baseline]
  Secondary measure of readiness to change/engage in pain self-management. 8 item questionnaire with range 0-48. Higher scores indicate more committed action/readiness.
Parental pain catastrophizing | At treatment admission and discharge, following intervention/control period
  Measure of parents' negative thoughts related to child's pain
Adult responses to child pain - protect subscale | At treatment admission and discharge, following intervention/control period
  Parental protective responses to child pain behaviors
Parental fear of pain questionnaire | At treatment admission and discharge, following intervention/control period
  Parent report of pain related fears/worries

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
THis is a very small, early phase RCT. There may be specific circumstances in which it would be appropriate to share our data. We welcome contact from investigators in the area of pediatric pain and would work to determine best sharing practices if relevant. All data would be de-identified.

REFERENCES:
- [Derived] Smith AM, Logan DE. Promoting readiness and engagement in pain rehabilitation for youth and families: Developing a pediatric telehealth motivational interviewing protocol. Paediatr Neonatal Pain. 2021 Oct 28;4(3):125-135. doi: 10.1002/pne2.12063. eCollection 2022 Sep. PMID 36188162